CLINICAL TRIAL: NCT02250599
Title: Multi-center, Randomized, Controlled, Open-label Study of Bevacizumab With Carboplatin and Paclitaxel Versus Carboplatin and Paclitaxel in Patients With Metastatic Nasopharyngeal Carcinoma
Brief Title: Efficacy and Safety of TC+AVASTIN Versus TC in Patients With Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML29153
Record Dates: First submitted 2014-08-26; First posted 2014-09-26 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Metastatic Nasopharyngeal Carcinoma; treatment
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma | interventions — Paclitaxel; Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carboplatin and paclitaxel (Active Comparator): carboplatin and paclitaxel :paclitaxel 175 mg/m2 IV and carboplatin AUC 6 IV on Day 1 of each 3-week cycle
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- AVASTIN and carboplatin and paclitaxel (Experimental): AVASTIN and carboplatin and paclitaxel: Bevacizumab(AVASTIN) 7.5 mg/kg intravenously (IV) infusion on Day 1 of each 3-week cycle; paclitaxel 175 mg/m2 IV and carboplatin AUC 6 IV on Day 1 of each 3-week cycle
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 175 mg/m2 IV Day 1 each 3-week cycle
Drug: Bevacizumab — Bevacizumab 7.5 mg/kg Day 1 each 3-week cycle
  Other Names: AVASTIN
  Arms: AVASTIN and carboplatin and paclitaxel
Drug: Carboplatin — Carboplatin AUC 6 IV Day 1 each 3-week cycle

SUMMARY:
The present study will be a randomized, control, multicenter phase II study of metastatic nasopharyngeal carcinoma (NPC) treated with evacizumab (AVASTIN,Roch) with paclitaxel and carboplatin regimen (TC+AVASTIN) or carboplatin/paclitaxel alone (TC). The population consists of metastatic nasopharyngeal carcinoma (NPC) that failed the radical radiotherapy or chemotherapy-naïve advanced NPC (stage IV). The effectiveness and side effects will be evaluated according to RECIST 1.1 and NCI-CTC AE V4.0.TEORTC QLQ-C30 and EORTC QLQ-H&N35 are used to measure PRO outcome for this study.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma is vastly more common in East Asia, especially China has a high incidence of it, and the number of new cases will account for more than 40% of the world total . The disease involved population maybe more than 4 million in the world. More than 2700-3000 new nasopharyngeal carcinoma patients will be diagnosed in SUN YAT-SEN university cancer center every year. It is most common in 40-50 years old adults and has been a top ten (10th) malignant tumor in Chinese male which threaten human health and social economy.

Chemotherapy is the standard treatment of the advanced nasopharyngeal carcinoma.Several other phase II study also confirmed the effectiveness of paclitaxel and carboplatin （TC） regimen in advanced NPC, so it maybe a simple right choice.

Increasing expression of VEGF in serum associated with poor prognosis in metastatic nasopharyngeal carcinoma. Agents that selectively target VEGF-A and its receptors have shown significant antitumor effects in xenograft models of nasopharyngeal. Studies demonstrated that bevacizumab（AVASTIN） administration with chemotherapy or chemoradiation is feasible in patients with nasopharyngeal cancer. Bevacizumab can be safely combined with a range of cytotoxic and other anticancer agents including TC regimen.

Evidence indicated a potential possibility that the TC+AVASTIN regimen may be superior than TC regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria for study entry:
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status 0~1
* Patients with a life expectancy>12 weeks
* Histologically proven NPC diagnosis
* Metastatic nasopharyngeal carcinoma with evidence of unsuitable for local treatment(in terms of some relevant therapy for anti-tumor like surgery, radiofrequency ablation, transcatheter arterial chemoembolization(TACE) and radiotherapy(except palliative radiotherapy for metastatic bone pain with appropriate radiation dosage without influence to the hemogram),etc.)
* Neoadjuvant or concurrent chemoradiotherapy was allowed, provided that the treatment was completed at least 3 months before the start of study drug treatment

  -≥1 measurable target based on RECIST criteria
* Adequate bone marrow, hepatic and renal function, defined as follows within 1 weeks prior to randomization
* Patients must sign study specific informed consent prior to registration
* Patient must have recovered (be >28 days post-surgery) from the effects of surgery, postoperative infection, and other complications before initial treatment with bevacizumab
* Systolic blood pressure ≤ 160 mmHg and diastolic pressure ≤ 90 mmHg within 7 days prior to randomization.

Exclusion Criteria:

* Prior systemic treatment for metastatic nasopharyngeal carcinoma
* Preparing for receiving local treatment for metastatic nasopharyngeal carcinoma (excluding palliative irradiation to release skeletal pain)
* Prior treatment with bevacizumab or other agents specifically targeting VEGF
* Patients with hemorrhage tendency including acute hemorrhage of digestive tract, nasal bleeding （not including nasal epistaxis), continuous hemorrhagic disease or Coagulation function disorder disease. Patients are using known NSAIDS to inhibit platelets.
* Patients with gross hemoptysis or hematemesis (defined as bright red blood of 1 teaspoon or more or frank clots within minimal or no phlegm per coughing episode) within 4 weeks prior to registration; patients with incidental blood mixed with phlegm are not excluded
* Patients receiving other experimental therapeutic cancer treatment
* Severe, active co-morbidity, defined as follows:

  i.--Unstable angina and/or congestive heart failure or vascular (e.g. aortic aneurysm requiring surgical repair or peripheral thrombosis) disease requiring hospitalization within the last 12 months, or other cardiac compromise (e.g. an inadequately controlled cardiac arrhythmia) that in the judgment of the investigator will preclude the safe administration of a study drug; Patient must not show sign of recent myocardial infarction or ischemia by the findings of S-T elevations of ≥ 2mm on an EKG ii.--History of arterial thromboembolic events, venous thromboembolism >NCI CTCAE Grade 3, transient ischemic attack (TIA), cerebral vascular accident (CVA), transmural myocardial infarction (MI), or hypertensive crisis or hypertensive encephalopathy iii.--History of ongoing bleeding diathesis, hemorrhagic disorder, or coagulopathy iv.--Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration v.--History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, or active GI bleeding within the last 6 months prior to registration; vi.--Esophageal varices, non-healing ulcer, non-healing wound, or bone fracture within the last 6 months prior to registration vii.--Active, untreated infection and/or acute bacterial or fungal infection uiring intravenous antibiotics at the time of registration viii.--Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; ix. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects x. - Minor surgical procedure including placement of a vascular access device, within 2 days of the first study treatment
* Patients currently (within 10 days of study enrollment) taking warfarin, heparin, daily treatment with aspirin (> 325 mg/day), or nonsteroidal anti-inflammatory medications known to inhibit platelet function; treatment with dipyramidole, ticlopidine, clopidogrel, or cilostazol
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception;
* Prior allergic reaction to the study drug(s) involved in this protocol
* Contraindication to Bevacizumab
* Patients has another cancer history （not NPC）within 5 years before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | 3 years

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
Overall response rate (ORR,CR+PR) | 3 years
  Identified by investigators and independent radiologic review (IRC) respectively
Disease control rate(DCR,CR+PR+SD) | 3 years
  Identified by investigators and IRC respectively
Health-related quality of life | 3 years
Number of Participants with Adverse Events | 3 years
Progression free survival(PFS) | 3 years
  Identified by IRC

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (8):
- China (8):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Department of Medical Oncology,Cancer Center of Sun Yat-Sen University, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan

REFERENCES:
- [Derived] Zhou T, Yang Y, Ma S, Lin L, Zhou T, Zhang C, Ding X, Wang R, Feng G, Chen Y, Xu R, Huang Y, Zhang L. Bevacizumab versus placebo in combination with paclitaxel and carboplatin as first-line treatment for recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase II trial. ESMO Open. 2021 Dec;6(6):100313. doi: 10.1016/j.esmoop.2021.100313. Epub 2021 Nov 24. PMID 34837744